CLINICAL TRIAL: NCT06716723
Title: Scrotal Surgery After Laparoscopic Donor Nephrectomy: a Population-based Matched Cohort Study
Brief Title: Scrotal Surgery After Laparoscopic Donor Nephrectomy
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025 0906 443 005; 148377 (Other Grant/Funding Number: Canadian Institutes of Health Research Foundation Grant)
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Scrotal Surgery; Living Kidney Donation; Nephrectomy,Kidney Donation
Keywords: living kidney donation; Scrotal surgery; cohort study; nephrectomy
MeSH Terms: interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- male kidney donors: Male kidney donors who had a laparoscopic nephrectomy between April 1, 2002 and March 31, 2023 at transplant centres in the province of Ontario, Canada. Each donor's nephrectomy date will serve as their cohort entry date.
  Interventions: Procedure: Nephrectomy
- male healthy nondonors: Before nephrectomy, living donors undergo rigorous health screening. We will select a similarly healthy segment of the general population using restriction and matching. We will randomly assign a cohort-entry date (simulated nephrectomy date) to all male citizens in Ontario, according to the distribution of cohort-entry dates among donors (between April 1, 2002 and March 31, 2023).
  We will identify baseline illnesses and measures of healthcare access using baseline records available before the cohort entry date. We will then restrict the sample to eligible nondonors without a recorded medical condition that could preclude donation. These restrictions will leave only a portion of citizens from the original sample as eligible nondonors.
  We will then match 10 eligible nondonors to each donor based on baseline characteristics that might be associated with the risk of scrotal surgery. Each nondonor can only be selected once.

INTERVENTIONS:
Procedure: Nephrectomy — Receipt of a laparoscopic nephrectomy for kidney donation
  Groups: male kidney donors

SUMMARY:
This study will examine whether laparoscopic nephrectomy is associated with a higher long-term risk of receiving scrotal surgery in male living kidney donors compared to male nondonors from the general population who have similar baseline health indicators. Both groups will be followed for many years.

DETAILED DESCRIPTION:
* Summary *

Background: It is underappreciated that some men who donate a kidney later experience unilateral scrotal pain and swelling on the same side of their nephrectomy. The condition can be assessed with an ultrasound, and some men undergo surgery for severe discomfort.

Methods: Using large provincial healthcare databases, we will conduct a retrospective cohort study of approximately 800 male kidney donors who will be matched in a 1:10 ratio with 8000 male nondonors of similar baseline health from the general population. Laparoscopic nephrectomies will have occurred between 2002 and 2023 in the province of Ontario, Canada, with follow-up through linked healthcare databases until March 2024. Donors and nondonors will be matched for age, date of cohort entry, residency (urban or rural), income (average neighbourhood income categorized into fifths), a history of vasectomy, and a history of inguinal hernia repair. The primary outcome will be a hospital admission with receipt of surgery to address a unilateral scrotal fluid collection, typically involving hydrocele excision. The secondary outcome will be receipt of a scrotal ultrasound.

Study outcome: The study will determine if laparoscopic nephrectomy is associated with a higher long-term risk of receiving scrotal surgery or a scrotal ultrasound in male living kidney donors compared to male nondonors with similar indicators of baseline health.

* Literature Review *

Over the last decade we have become aware of reports suggesting that some male donors experience unilateral testicular pain and scrotal swelling after donation on the same side of their nephrectomy. Upon review, we identified over 10 studies that have described this outcome. The proportion of affected male donors ranged from 2% to 55%. No study included a comparison group of nondonors, and most studies only followed donors for a short period after nephrectomy. Some studies reported that testicular pain was more common after laparoscopic than open surgery. The pain was described as dull, aching, and heavy in nature, starting in the week following nephrectomy. Some studies, but not others, report that testicular pain was more common after a left-sided versus right-sided nephrectomy, where, due to anatomy, the gonadal vein is divided in a left nephrectomy but may be spared in a right nephrectomy. There are several treatment options for testicular pain, including reports of some men undergoing scrotal surgery to address a hydrocele on the same side as their donated kidney.

* Research location *

The study will be conducted at ICES (ices.on.ca), an independent, non-profit research institute whose legal status under Ontario's health information privacy law allows it to collect and analyze health care and demographic data without consent for health system evaluation and improvement. The use of data in this project is authorized under section 45 of Ontario's Personal Health Information Protection Act, which does not require review by a Research Ethics Board.

Information will be obtained from several linked databases in Ontario such as, the Trillium Gift of Life Network, Ontario's Registered Persons Database, and the Ontario Health Insurance Plan, and from the Canadian Institute for Health Information the Discharge Abstract Database, National Ambulatory Care Reporting System and Same Day Surgery. In Ontario, the Canadian Classification of Health Interventions system to record procedures in healthcare databases was adopted on April 1, 2002, and this date will serve as the start of our accrual period. We expect the data to be complete for virtually all variables to be used in this study. This is a retrospective cohort study for which all study data is already available in administrative healthcare databases at ICES. As a recommended research practice, we are publicly documenting the study description, design and statistical analysis plan on clinicaltrials.gov. before analyzing the study outcomes.

* Statistical analysis plan *

Baseline characteristics: Continuous variables will be presented as mean (standard deviation) or median (interquartile range [IQR]), as appropriate, and categorical variables as frequency (percentage). Due to our large expected cohort size and the influence of sample size on statistical testing, the characteristics of donors and nondonors at the time of cohort entry will be compared prior to and after matching using standardized mean differences, where a value >0.10 is considered meaningfully different. Characteristics specific to the donors will also be reported (e.g., pre-nephrectomy kidney function, their relationship to the recipient, the number of years the surgeon who performed their nephrectomy was in practice).

Period of observation: After cohort entry, a person's follow-up time will be censored at the time of developing the relevant study outcome (i.e., time to first event), death, emigration from the province, or the end of the study's observation period (March 31, 2024).

Assessing risk of the primary and secondary outcome: The association between laparoscopic donor nephrectomy and a hospital admission with scrotal surgery will be assessed using hazard ratios and their 95% confidence intervals, estimated using Cox proportional hazards regression with robust variance estimation accounting for the correlation within matched sets. The proportional hazards assumption will be assessed using the Kolmogorov-type supremum test on 1000 simulated patterns. If the assumption is violated, instead of a hazard ratio, a stratified log-rank test will be used to test significance of the outcome and the difference of restricted mean survival time at 20 years with its 95% confidence interval will be presented.

Main additional analyses:

(i) We will perform the primary outcome analysis restricting the code set only to hydrocele repair.

(ii) Our primary focus is to better understand the outcomes following laparoscopic donor nephrectomy, which currently is the preferred method for this procedure. However, over 250 open nephrectomies were also performed in Ontario during the study period. Some studies suggest that scrotal symptoms may be more common after laparoscopic procedures compared to open ones, while other studies do not support this claim. To investigate this, we will add a group of donors who underwent open procedures during the study period, assembled in a similar fashion to those who had laparoscopic procedures. We will employ inverse probability of treatment weighting based on propensity scores to balance the baseline characteristics of the donors who had nephrectomies via laparoscopic procedures (one group) and open procedures (the other group). Donors who had open procedures will be weighted using the average treatment effect in the treated weights, defined as propensity score divided by (1 - propensity score). Donors who received laparoscopic procedures will have a weight of 1. This approach is expected to generate a weighted pseudo-sample of donors who underwent open procedures, with a distribution of measured baseline characteristics resembling that of donors who had laparoscopic procedures. We will account for the weighting in all comparative analyses, with hazard ratios estimated using Cox proportional hazards regression and 95% confidence intervals created using a variance estimate obtained from bootstrapping. Our primary outcome will be receipt of scrotal surgery, while our secondary outcome will be receipt of a scrotal ultrasound.

(iii) If we can reliably ascertain the side of nephrectomy in our data sources, we will compare the outcomes of left vs. right nephrectomy amongst those who received a laparoscopic nephrectomy. This will be done in the same manner as for open vs. laparoscopic nephrectomy. Some studies, but not others, report that scrotal symptoms are more common after a left-sided versus right-sided nephrectomy, where, due to anatomy, the gonadal vein is divided in a left nephrectomy but may be spared in a right nephrectomy.

Other additional analyses

(iv) We will conduct the primary and secondary outcome analysis for other prespecified subgroups of men according to age, income, year of cohort entry, and a history of vasectomy prior to cohort entry (yes or no), and if the number of events allow for meaningful analysis, rural residence and a prior history of inguinal hernia repair. We expect no significant difference in the hazard ratio between these subgroups. Rather, they will be examined for general consistency of any donation-attributable observed effect across subgroups.

(v) We will analyze the characteristics associated with our primary and secondary outcomes separately for donors and nondonors using Cox proportional hazards regression. The characteristics under consideration and assessed at cohort entry include age, income, rural residence, year of cohort entry, a prior history of vasectomy, and a prior history of inguinal hernia repair. In nondonors, an older (vs. younger) age at cohort entry may associate with a higher risk of developing the outcomes in follow-up, whereas this association may not hold true for donors. Rather, in donors, outcomes caused by nephrectomy may be minimally associated with age at cohort entry.

Descriptive analyses and graphs

(i) Outcomes will be described as incidence rates per 1000 person-years, and as the cumulative incidence during follow-up (obtained using the Aalen-Johansen estimator, treating death as a competing event, with donors and nondonors compared visually with graphical curves and at landmark timepoints).

(ii) Characteristics of the primary outcome amongst donors will be described, such as when the scrotal surgeries were performed after nephrectomy, whether they were done under general anesthesia, whether they required a hospital overnight stay, and whether they were performed by a different surgeon than the one who performed their nephrectomy. Similarly, we will examine the characteristics of the secondary outcome amongst donors, such as the type of physician who ordered the scrotal ultrasound and when it was performed after nephrectomy.

P values (significance testing) and confidence intervals: We will perform hierarchical statistical tests to assess our hypotheses in the pre-defined order described below. The 2-sided significance level will be 0.05 for each tested hypothesis. After a non-significant test no further significance testing will be performed and no further P values will be reported. All estimates (with and without P values) will be reported as point estimates with 95% confidence intervals. We acknowledge the interval widths of the estimates without P values are not adjusted for multiple testing and that those inferences may not be reproducible. The order:

(i) the primary outcome (scrotal surgery) in donors vs. nondonors (ii) the secondary outcome (scrotal ultrasound) in donors vs. nondonors (iii) hydrocele surgery (codes within the primary outcome) in donors vs. nondonors (iv) primary outcome in donors who underwent a laparoscopic vs. open procedure (v) secondary outcome in donors who underwent a laparoscopic vs. open procedure (vi) [if data on laterality is available] primary outcome in donors who underwent a left vs. right laparoscopic nephrectomy (vii) [if data on laterality is available] secondary outcome in donors who underwent a left vs. right laparoscopic nephrectomy

Statistical power: We are restricted to using information available in our datasets and have not performed power calculations to determine the sample size needed to detect a given effect with adequate statistical power. Instead, we will present 95% confidence intervals with our point estimates to suggest the range in which the true parameter may fall. There are now over 10 studies describing testicular pain and/or scrotal swelling in donors, with a range of 2% to 55% of donors effected. This study will produce the first population-based estimates of donation-attributable absolute and relative risks with 95% confidence intervals of this potentially important complication.

ELIGIBILITY:
* Donors *

  * Male persons who received a laparoscopic nephrectomy in Ontario, Canada between April 1, 2002, and March 31, 2023 are eligible to enter the study.
  * We will exclude any person with data errors in their database records (such as missing or invalid age; we expect to exclude very few persons for these reasons). Data errors also include evidence of prior dialysis or a prior solid organ transplant, as such persons are not eligible to become a donor.
  * We will exclude any person who was not a permanent Ontario resident (i.e., they live outside of Ontario, and only came to Ontario to donate a kidney to their intended recipient). This will include anyone who is not eligible for the Ontario Health Insurance Plan, anyone whose date of last contact in our databases is less than 4 months after the cohort entry date, and any person without a physician visit in the last 1-year.
  * We will exclude any person who is <18 years of age on the date of nephrectomy (as only under exceptional circumstances should a person less than 18 be approved for living donation).
  * We will exclude any person who, before donation, received a scrotal ultrasound or a scrotal procedure other than a vasectomy.
* Non-donors *

  * Before nephrectomy, living donors undergo rigorous health screening. We will select a similarly healthy segment of the general population using restriction and matching.
  * We will randomly assign a cohort-entry date (simulated nephrectomy date) to all male persons who were citizens in Ontario, according to the distribution of cohort-entry dates among donors (April 1, 2002, to March 31, 2023).
  * We will exclude any person with data errors in their database records (such as missing or invalid age).
  * We will exclude any person who was not a permanent Ontario resident. This will include anyone who is not eligible for the Ontario Health Insurance Plan, and anyone whose date of last contact in our databases is less than 4 months after the cohort entry date
  * We will exclude any person who is <18 years of age on the cohort entry date
  * We will identify baseline illnesses and measures of healthcare access from historic records preceding the cohort entry date. We will then restrict the sample of eligible nondonors to persons without a recorded medical condition that could preclude donation. Such recorded medical conditions will include a hospitalization for mental illness in the prior year; an intensive care unit admission in the prior year; a hospitalization for palliative care services in the prior year; multiple hospital admissions in the prior year; high comorbidity (as assessed by the Charlson comorbidity index and adjusted clinical group scores); receipt of home oxygen therapy; residence at a long-term care facility; dementia; any record of prior nephrology consultation or kidney disease (including receipt of dialysis, a kidney biopsy, or a kidney procedure such as a partial or complete nephrectomy); previous solid organ transplant; disorders of the kidneys, ureters, or bladder; any record of cardiovascular disease (congestive heart failure, cardiovascular procedures, myocardial infarction, peripheral vascular disease, abdominal aortic aneurysm repair, ischemic stroke); hypertension in individuals <50 years of age (persons with this condition are not accepted as donors in Ontario); any record of obstructive sleep apnea; any cancer diagnosis; any liver disease or cirrhosis; diabetes; any serious infection (hepatitis, HIV, infective endocarditis); any record of autoimmune rheumatic conditions (such as rheumatoid arthritis or systemic lupus erythematosus); and any record of alcoholism.
  * We will exclude any person who, before cohort entry, received a scrotal ultrasound or a scrotal procedure other than a vasectomy.
  * To ensure the nondonors have the same opportunity as donors to obtain health care services from physicians, we will exclude nondonors who had no evidence of a family physician visit in the 2 years prior to index. We will also exclude nondonors with more than 4 family physician visits in the 2 years prior to index, as this could suggest they have an active health issue that needs attention before they would proceed to donate.
* Matching *

We will then match each donor to 10 eligible nondonors based on baseline characteristics that might be associated with the risk of scrotal surgery, specifically the age at the time of cohort entry (± 1 years), since amongst adults, as men age they are more likely to have hydroceles; the cohort entry date (± 3 years), to account for any era effects; urban or rural residence (population ≥ 10,000 or < 10,000), as a rural residence is associated with less access to care and worse outcomes; income (categorized into fifths of average neighborhood income), since lower income is associated with less access to care and worse outcomes; a prior history of vasectomy, and a prior history of inguinal hernia repair, as each procedure on occasion leads to chronic testicular pain. Each nondonor can only be selected once.

Ages: 18 Years to 106 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male kidney donors who underwent laparoscopic nephrectomy matched to male nondonors from the general population with similar indicators of baseline health.
Sampling Method: Non-Probability Sample
Enrollment: 9878 (Actual)
Dates: Start 2002-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Scrotal Surgery | Donors and their matched non-donors will enter the cohort between April 1, 2002 and March 31, 2023, and will be followed until study outcome (first event), death, emigration from the province, or the end of the observation period (March 31, 2024).
  Hospital admission and receipt of surgery for a unilateral scrotal fluid collection such as hydrocele excision. To be confident in outcome ascertainment, evidence of both a surgeon-fee-for-service code and a hospital-based procedural code will be required, with each recorded in separate healthcare databases by different personnel.

SECONDARY OUTCOMES:
Scrotal Ultrasound | Donors and their matched non-donors will enter the cohort between April 1, 2002 and March 31, 2023, and will be followed until until study outcome, death, emigration from the province, or the end of the observation period (March 31, 2024).
  Receipt of a scrotal ultrasound. This test is typically ordered to evaluate a person with ongoing pain or swelling in their scrotum or testis.

CONTACTS AND LOCATIONS:
Locations (1):
- ICES, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The dataset from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). The full dataset creation plan and underlying analytic code are available from the authors upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Derived] Garg AX, McArthur E, Sontrop JM, Boudville N, Connaughton DM, Cuerden MS, Feldman LS, Lam NN, Lentine KL, Nguan C, Parikh CR, Segev DL, Sener A, Smith G, Wang C, Weir MA, Yohanna S, Young A, Naylor KL. Risk for Scrotal Surgery After Laparoscopic Donor Nephrectomy : A Population-Based Cohort Study. Ann Intern Med. 2026 Jan;179(1):23-31. doi: 10.7326/ANNALS-25-02257. Epub 2025 Nov 11. PMID 41213151